CLINICAL TRIAL: NCT05537961
Title: Impact of Mindfulness Training on Adolescent Well-Being and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Cambron, Assistant Professor, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00122449
Record Dates: First submitted 2022-08-18; First posted 2022-09-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Substance Use; Mindfulness; Psychological Well-being
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Weekly mindfulness instruction embedded in classroom setting
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement
- No Intervention (No Intervention): Classroom setting completed as usual

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — Mindfulness instruction incorporated in classroom-based curriculum
  Arms: Mindfulness

SUMMARY:
There is a broad consensus that preventing or delaying initiation of adolescent alcohol, tobacco, and other drug (ATOD) use can substantially improve both short- and long-term adolescent health. Despite the existence of effective prevention programs, adolescent ATOD use continues to be a substantial issue. Continued research on preventive interventions is needed. School-based mindfulness-based interventions (MBIs) have been shown to be feasible and effective at improving adolescent psychological well-being. Evidence from both quasi-experimental studies and randomized controlled trials suggests that incorporating MBIs into school-settings can lower levels of anxiety, depression, and stress, while improving capacity for emotional regulation. Greater mindfulness also been linked to reduced adolescent ATOD use via observational studies. There are strong theoretical reasons to believe that MBIs delivered in school settings can prevent or reduce ATOD use among youth. In particular, MBIs have been shown to improve psychological well-being among youth via multiple mechanisms also relevant for adolescent ATOD use. These mechanisms include enhanced attentional control, negative emotion regulation, promotion of positive emotion generation, and increased feelings of connectedness. Despite these connections, school-based MBIs are yet to demonstrate the ability to prevent or reduce adolescent ATOD use.

The current study will examine psychological well-being and ATOD use among approximately 80 participants in a quasi-experimental, school-based MBI. In early 2022, approximately 40 high school seniors were provided with one semester of a weekly, classroom-based MBI embedded into their Social Studies curriculum; approximately 40 high school seniors participated in the standard curriculum. The intervention group was provided with an adaptation of Mindfulness-Oriented Recovery Enhancement (MORE). MORE is an evidence-based therapeutic program that integrates mindfulness, cognitive-behavioral therapy, and positive psychology to treat addiction and enhance well-being. MORE has been shown to produce therapeutic benefits in the treatment of alcohol, tobacco, and other drug addiction in adult populations, but is yet to be tested as a preventive intervention for youth. Follow up data collection is planned for spring 2023 to assess psychological well-being, ATOD use, and proposed therapeutic mechanisms pre-intervention, post-intervention, and at 9-month follow up.

DETAILED DESCRIPTION:
There is a broad consensus that preventing or delaying initiation of adolescent alcohol, tobacco, and other drug (ATOD) use can substantially improve both short- and long-term adolescent health. Despite the existence of effective prevention programs, adolescent ATOD use continues to be a substantial issue. Continued research on preventive interventions is needed. School-based mindfulness-based interventions (MBIs) have been shown to be feasible and effective at improving adolescent psychological well-being. Evidence from both quasi-experimental studies and randomized controlled trials suggests that incorporating MBIs into school-settings can lower levels of anxiety, depression, and stress, while improving capacity for emotional regulation. Greater mindfulness also been linked to reduced adolescent ATOD use via observational studies. There are strong theoretical reasons to believe that MBIs delivered in school settings can prevent or reduce ATOD use among youth. In particular, MBIs have been shown to improve psychological well-being among youth via multiple mechanisms also relevant for adolescent ATOD use. These mechanisms include enhanced attentional control, negative emotion regulation, promotion of positive emotion generation, and increased feelings of connectedness. Despite these connections, school-based MBIs are yet to demonstrate the ability to prevent or reduce adolescent ATOD use.

The current study will examine psychological well-being and ATOD use among approximately 80 participants in a quasi-experimental, school-based MBI. In early 2022, approximately 40 high school seniors were provided with one semester of a weekly, classroom-based MBI embedded into their Social Studies curriculum; approximately 40 high school seniors participated in the standard curriculum. The intervention group was provided with an adaptation of Mindfulness-Oriented Recovery Enhancement (MORE). MORE is an evidence-based therapeutic program that integrates mindfulness, cognitive-behavioral therapy, and positive psychology to treat addiction and enhance well-being. MORE has been shown to produce therapeutic benefits in the treatment of alcohol, tobacco, and other drug addiction in adult populations, but is yet to be tested as a preventive intervention for youth. Follow up data collection is planned for spring 2023 to assess psychological well-being, ATOD use, and proposed therapeutic mechanisms pre-intervention, post-intervention, and at 9-month follow up. Trajectories of change will be assessed to test the following three aims.

Aim 1 is to examine the impact of MORE on changes in students' psychological well-being (i.e., anxiety, depression, stress) and ATOD use relative to a standard curriculum. The investigators hypothesize that MORE will improve psychological well-being and reduce ATOD use, relative to the standard curriculum.

Aim 2 is to examine the impact of MORE on changes in students' attentional control (i.e., mindfulness), negative emotion regulation (i.e., positive reappraisal), positive emotion generation (i.e., savoring), and feelings of connectedness (i.e., self-transcendence) relative to a standard curriculum. The investigators hypothesize that MORE will improve attentional control, negative emotion regulation, and positive emotion generation, as well as increasing feelings of connectedness, relative to a standard curriculum.

Aim 3 is to examine the extent to which MORE encourages improved psychological well-being and reduced ATOD use via the therapeutic mechanisms identified in Aim 2 (attentional control, negative emotion regulation, positive emotion generation, and feelings of connectedness). The investigators hypothesize that the relationship between MORE and positive outcomes will be mediated by the proposed therapeutic mechanisms.

Hypothesis: Results of the current study will provide important information to advance the fields of both ATOD prevention and school-based MBIs. Additionally, results of this study will be of wide interest to school administrators, school counselors, and clinicians working to prevent adolescent substance use. Successful completion of this study will lead to multiple publications. Additionally, results of this study will provide essential pilot data to inform further testing of MORE for adolescents via randomized controlled trials and support multiple possible grant submissions. While MBIs have become a common part of substance abuse treatment among adults, school-based MBIs for ATOD prevention lack sufficient evidence and are yet to be regularly incorporated into standard prevention efforts.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a high school senior in two specific classes at Judge Memorial High School during Spring 2022

Exclusion Criteria:

* Not enrolled as a high school senior in two specific classes at Judge Memorial High School during Spring 2022

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Youth Risk Behavior Surveillance System: Substance use | change in each measure across 9 months
  alcohol, tobacco, and other drug use as measured by the Youth Risk Behavior Surveillance System. Items are measured as any use on both lifetime and past 30 days.
Youth Risk Behavior Surveillance System: Suicide ideation | change in each measure across 9 months
  suicide ideation and attempts as measured by the Youth Risk Behavior Surveillance System. Suicide ideation is measured as any ideation in the past 12 months and attempts are measured as the count of attempts in the past 12 months.
Pediatric Patient Reported Outcomes Measurement Information System (PROMIS) | change in each measure across 9 months
  positive affect, life satisfaction, meaning and purpose, anxiety, depressive symptoms as measured by the pediatric PROMIS. For each scale, higher scores indicate higher levels of the name of the scale. Items on each scale are summed and T scores with a mean of 50 and standard deviation of 10 are calculated.
Child Acceptance and Mindfulness Measure | change in each measure across 9 months
  Mindfulness as measured by the child acceptance and mindfulness measure (CAMM). The CAMM is scored from 0 to 40 with higher scores indicating higher levels of mindfulness
Cognitive Emotion Regulation Questionnaire | change in each measure across 9 months
  Positive reappraisal as measured by the Cognitive Emotion Regulation Questionnaire (CERQ). The CERQ is scored from 1 to 7 with higher scores indicating higher levels of emotion regulation.
Nondual Awareness Dimensional Assessment | change in each measure across 9 months
  Transcendental experiences as measured by the Nondual Awareness Dimensional Assessment (NADA). Higher scores indicate greater nondual awareness trait scored from 0 to 12 and nondual awareness states scores from 0 to 40
Toronto Mindfulness Scale | change in each measure across 9 months
  Mindfulness as measured by the Toronto Mindfulness Scale. Higher scores indicate higher degree of state mindfulness. Scores range from 0 to 24 on the curiosity subscale and from 0 to 28 on the decentering subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cambron, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No